CLINICAL TRIAL: NCT05248282
Title: A Single-Center, Retrospective, Blinded Validation Study to Investigate the Prognostic Value of the Prostatype Test System (PrTS) in Prostate Cancer Patients in China
Brief Title: Clinical Validation of the Prognostic Value of the PrTS on Prostate Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Prostatype Genomics AB (Unknown); GloriousMed Clinical Laboratory (Shanghai) Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Hongqian Guo, Director of Urology Department, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: IUNU-PC-107
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prostate Cancer is the most common type of cancer among men in many countries. However current clinical tools have limited prediction accuracy to choose the optimal treatment for the individual patient, as prostate cancer risk assessment is a critical aspect of treatment decision-making. A substantial proportion of patients are undergoing over-treatment such as radical treatment, which is often associated with negative physical and psychological side effects, dramatically affecting quality of life in a negative way. Moreover, the patients that are under-treated will face higher cancer mortality risks, which brings more concerns for patients and doctors. Prostatype composes a one-step 4-plex quantitative reverse transcription polymerase chain reaction kit, a database based on authenic patients information and a score system (P-score), intended to measure gene expression levels of three biomarkers: IGFBP3, F3 and VGLL3. Genetic values combined with clinical parameters in the CPMA and P-score are aiming to estimate the aggressiveness of prostate tumor for a newly diagnosed prostate cancer patient. This is a single-center, retrospective, blinded validation study aim to investigate the prognostic performance of the Prostatype test system.

ELIGIBILITY:
Inclusion Criteria:

* Non-metastatic prostate adenocarcinoma confirmed by histopathology after taking core needle biopsy
* Regular visits, treatment and laboratory tests were conducted in the past
* There is biopsy materials at the time of diagnosis (without staining FFPE)
* The total area of tumor tissue shall be 25-30 mm2, and the proportion of tumor cells after tumor cell enrichment is at least 50%
* Complete records of relevant clinical follow-up information

Exclusion Criteria:

* Biopsy tissue is not available, or FFPE does not meet the screening requirements of study samples
* Relevent clinical parameters of the patients are not available
* Treatment methods are not available
* Age of diagnosis < 50 years
* Age of diagnosis > 100 years
* Total tumor length < 2 mm
* The patient died of an accident, homicide or suicide

Ages: 50 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men diagnosed with non-metastatic prostate cancer
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
prostate cancer-specific mortality | up to 36 months
  To verify that the prediction performance of risk stratification model (P-score) in the Chinese population is superior to that of the current European Society of Urology (EAU) risk stratification standard with regard to prostate cancer-specific mortality

SECONDARY OUTCOMES:
metastasis-free survival | up to 36 months
  To investigate that the prediction performance of risk stratification model (P-score) in the Chinese population is superior to that of the current European Society of Urology (EAU) risk stratification standard with regard to metastasis free survival
Prognostic value of the three gene-signature in P-score | up to 36 months
  To verify the prognostic value of the three gene-signature (IGFBP3, F3 and VGLL3) in Chinese population, explore their association with prostate cancer-specific mortality and metastasis free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, Nanjing, Jiangsu, China